CLINICAL TRIAL: NCT03779802
Title: Comparison of the Acute Hemodynamic Effect of Three Modes of Stimulation in Cardiac Resynchronization.
Brief Title: Prospective Multicentric Study Comparing the Acute Hemodynamic Effect of Three Modes of Stimulation in Cardiac Resynchronization Therapy Recipients
Acronym: 3 STIM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: With the current health situation, we do not anticipate a significant resumption of recruitment for several months.
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/10
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure; Cardiac Resynchronization Therapy
Keywords: Cardiac Resynchronization Therapy; Atrioventricular delay optimization; Multipoint pacing; Negative atrioventricular hysteresis; Non invasive hemodynamic optimization; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Defibrillators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRT device (Experimental): Patients implanted with a CRT device who will undergo a non-invasive hemodynamic evaluation of different pacing modes
  Interventions: Other: Device programming of ABBOTT CRT pacemaker or defibrillator

INTERVENTIONS:
Other: Device programming of ABBOTT CRT pacemaker or defibrillator — Comparison of the acute hemodynamic effect of three modes of stimulation in ABBOTT CRT devices (Biventricular, SyncAV and MPP modes) by using the Finapress® NOVA method to assess the highest systolic blood pressure (SBP) during the programming session Comparison of the acute hemodynamic effect of three modes of stimulation in ABBOTT CRT devices (Biventricular, SyncAV and MPP modes) by using the Finapress® NOVA method to assess the highest systolic blood pressure (SBP) during the programming session.

SUMMARY:
Cardiac Resynchronization Therapy (CRT) is an established treatment for patients with systolic heart failure and bundle branch block, improving functional capacity, quality of life and reducing morbi-mortality.

Adjusting atrio-ventricular (AV) delay, vector optimization and choice of different modes of stimulation can influence the acute hemodynamical consequences of CRT but also its medium-term and long-term clinical and echocardiographic effects.

The aim of the present prospective study is to investigate whether the different stimulation modes lead to different acute hemodynamic response, by evaluating the highest systolic pressure using the Finapress ® method.

DETAILED DESCRIPTION:
This study is a non-randomized, prospective, interventional, multicentric study.

Patients implanted with an Abbott ® CRT pacemaker or defibrillator since less than 3 months are eligible for the study.

Recruited patients will be submitted to a non-invasive evaluation of different pacing modes. This will be performed using the Finapress NOVA device, which records blood pressure with a digital cuff. The peak of blood pressure will correspond to the optimal device settings

Three modes of stimulation of ABBOTT CRT devices will be compared:

* Classical bi-ventricular pacing mode at nominal value and with AV delay optimization
* SyncAV mode at nominal value or with left ventricular preexcitation optimization
* Multipoint Pacing (MPP) mode, alone or in combination with SyncAV mode This is an acute evaluation study without scheduled follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18
* Implantation of a CRT (CRT-P or CRT-D) less than 3 months before inclusion
* MPP and SyncAV-enabled ABBOTT Quadripolar CRT pacing system
* Patient who had signed an informed consent and is willing to comply with study requirements
* De novo implantation
* Patient covered by national healthcare insurance

Exclusion Criteria:

* Permanent/persistant atrial fibrillation/ supra-ventricular tachycardia
* Pacing indication for 2nd or 3rd degree AV block
* Upgrading from non-CRT system
* Pregnant or breastfeeding women
* Adult under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-04-18 (Actual); Study Completion 2020-04-18 (Actual)

PRIMARY OUTCOMES:
Hemodynamic response | day 0
  Highest Systolic Blood Pressure (SBP) obtained by optimization of the mode of stimulation

SECONDARY OUTCOMES:
Other hemodynamical response | day 0
  Cardiac output
Other hemodynamical response | day 0
  Systolic ejection volume
Other hemodynamical response | day 0
  dP/dT

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan MD MOUBARAK, Principal Investigator — CMC Ambroise Paré
Locations (3):
- France (3):
  - Gehm Site D'Eaubonne, Eaubonne, Val-d'Oise
  - Cmc Ambroise Pare, Neuilly-sur-Seine
  - CHU Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferchaud V, Garcia R, Bidegain N, Degand B, Milliez P, Pezel T, Moubarak G. Non-invasive hemodynamic determination of patient-specific optimal pacing mode in cardiac resynchronization therapy. J Interv Card Electrophysiol. 2021 Nov;62(2):347-356. doi: 10.1007/s10840-020-00908-6. Epub 2020 Oct 30. PMID 33128179